CLINICAL TRIAL: NCT02408185
Title: Pharmacokinetics and Pharmacodynamics of Colistin in Critically Ill Patients With Severe Infections for Dose Optimization Study
Brief Title: Optimization Dose Study on Pharmacokinetics and Pharmacodynamics of Colistin in Critically Ill Patients
Acronym: COLPHAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MagicBullet/COLPHAR
Record Dates: First submitted 2015-03-23; First posted 2015-04-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Critical Illness
Keywords: infections; multidrug resistant Gram negative bacteria (MDR-GNB); Skin infections; Pneumonia; Bacteriemia; Nosocomial infections
MeSH Terms: conditions — Critical Illness; Infections; Cellulitis; Pneumonia; Cross Infection | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colistin 6 million units + 240mg/8h (Experimental): Loading dose of 6 million units of colistin+ 240mg/8h maintenance
  Interventions: Drug: Colistin 6 million units + 240mg/8h
- Colistin 6 million units + 360mg/12h (Experimental): Loading dose of 6 million units of colistin+ 360mg/12h maintenance
  Interventions: Drug: Colistin 6 million units + 360mg/12h

INTERVENTIONS:
Drug: Colistin 6 million units + 240mg/8h — 240 mg of colistin methanesulfonate (CMS) every 8 hours, 3 million units (MU); 90 mg colistin base activity, (CBA)
  Other Names: colistin methanesulfonate (CMS); colistin base activity (CBA)
  Arms: Colistin 6 million units + 240mg/8h
Drug: Colistin 6 million units + 360mg/12h — 360 mg CMS every 12 hours (4.5 MU; 135 mg CBA)
  Other Names: colistin methanesulfonate (CMS); colistin base activity (CBA)
  Arms: Colistin 6 million units + 360mg/12h

SUMMARY:
Phase II clinical trial, open-labelled, prospective and single-center study directed to obtain blood samples in experimental detailed conditions in order to compare and optimize the dose of colistin in critically ill patients suffering from infections on which the indication of colistin would be accepted according to normal local protocols for severe infections treatment.

ELIGIBILITY:
Inclusion Criteria:

* More than 60 Kg of weigh
* Patients with directed treatment with colistin as the recommended antimicrobial treatment protocols in the hospital to treat some of the following serious infections caused by carbapenems resistant A. baumannii: (i) bacteremia; (ii) nosocomial pneumonia or (iii) infection of skin and soft tissue (cellulitis, abscesses or infected ulcers).
* Written informed consent form.

Exclusion Criteria:

* Refractory shock or other illness with an expectative of life ˂ 48 hours after the recruitment;
* Patient declared not to resuscitation maneuvers;
* Suspicion or demonstration of endocarditis, osteomyelitis, or meningitis;
* Known hypersensitivity to polymyxins;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile; Cmax (maximum reach concentration)/ MIC( Minimum inhibitory concentration) >10 | Day 1 and day 3 after treatment
  Plasma concentration will be measured for pharmacokinetic and pharmacodynamic profile the samples were drawn at 60, 120, 180, 240, 360, and 480 min after the end of the loading dose infusion and in patients of the group B, two more samples are taken at 600 and 720 min after the loading dose. Main pharmacokinetic parameters will be Cmax (maximum reach concentration)/ MIC(Minimum inhibitory concentration)>10

SECONDARY OUTCOMES:
Number of drug adverse reactions | 21 days of follow-up
  All study drug related adverse reactions will be gathered and communicated.
Pharmacodynamic profile ("Monte-Carlo simulation" (statistical methodology) with MIC (Minimum inhibitory concentration) 50 y MIC (Minimum inhibitory concentration) 90 from samples isolation) | Day 1 and day 3 after treatment
  "Monte-Carlo simulation" (statistical methodology) with MIC (Minimum inhibitory concentration) 50 y MIC (Minimum inhibitory concentration) 90 from samples isolation

CONTACTS AND LOCATIONS:
Overall Officials: M. Eugenia Pachón, BD-PhD, Principal Investigator — Instituto de Biomedicina de Sevilla (IBIS); José Miguel Cisneros, MD-PhD, Study Chair — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No